CLINICAL TRIAL: NCT06218472
Title: Assessment of the Impact of Early Treatment for Anorexia Nervosa in a Day Hospital on Food Symptomatology, the Outcome of Young Patients, and the Family Experience
Acronym: EVA-FAM
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231594; 2023-A02047-38 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-01-08; First posted 2024-01-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; Family-based treatment; Day hospital; Early intervention; Parental experience
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Day hospital patient: Acceptance of the DH program (DH group): scheduling of 10 to 12 sessions over 12 weeks during a program session, followed by a reassessment at the end of the program. Outpatient follow-up thereafter.
  Interventions: Other: Day Hospital Treatment
- Outpatient: Refusal or inability to participate in the DH program: multidisciplinary follow-up "as usual" within the service (outpatient group).
  Interventions: Other: Multidisciplinary follow-up "as usual" within the service
- Parents
  Interventions: Other: Conduct semi-structured qualitative interviews

INTERVENTIONS:
Other: Day Hospital Treatment — Scheduling of 12 half-day sessions per week, alternating between sessions with only the patients or involving the entire family. Close medical monitoring and multidisciplinary interventions during sessions (pediatrician, psychiatrist, dietitian, recovered former patients...).
  Other Names: Family based treatment
  Groups: Day hospital patient
Other: Multidisciplinary follow-up "as usual" within the service — Multidisciplinary follow-up "as usual" within the service
  Groups: Outpatient
Other: Conduct semi-structured qualitative interviews — Conduct semi-structured qualitative interviews
  Groups: Parents

SUMMARY:
During the management of chronic illnesses, the day hospital (DH) serves as a brief and effective alternative to traditional hospitalization, offering access to multidisciplinary care. Indeed, patients can benefit from a range of therapeutic tools provided by a multidisciplinary care team while remaining in their living environment. Numerous structures exist for the management of eating disorders, but primarily for severe cases, often following hospitalization, before transitioning to outpatient care. There is no alternative for the initial management of these patients.

The DH for the evaluation and early intervention in recent forms of anorexia nervosa at Maison de Solenn serves as a rapid entry point to specialized care. It allows for a thorough assessment and sustained management of eating disorders. Our hypothesis is that a multidisciplinary, intensive, and early intervention for patients with anorexia nervosa and their families in a day hospital would improve the short, medium, and long-term prognosis of the disease compared to conventional multidisciplinary outpatient care. It would also enhance the family's experience of this pathology and their coping skills.

DETAILED DESCRIPTION:
The patients recruited will come from the active consultation file of the inclusion center (spontaneous consultations, referrals from healthcare professionals, etc.), whether they have had an initial consultation or not. All patients admitted to day hospital during the study period who meet the inclusion criteria will be considered. A first evaluation consultation for mental anorexia will be conducted for all patients, including a somatic and psychological assessment, as well as a consultation with a dietitian. If eligible, the patient and their family will be offered participation in day hospital (for the next session or the following one, depending on availability). In case of refusal, regardless of the reason (parents' availability, excessive distance from home, lack of motivation, etc.), patients will receive regular care in outpatient consultations. For the qualitative study, parents participating in day hospital for their adolescent will be offered inclusion in this research protocol.

The inclusion of young patients will take place over two calendar years (24 consecutive months) for the characterization of the active file. The study will continue for 5 years after the inclusion of the last patient in the study to investigate the outcome. In total, data collection for this research will last a maximum of 84 months (24 months of recruitment and a 5-year follow-up).

Visit 1 - Inclusion: collection of non-oppositions, initial clinical evaluation, then proposal to participate in the day hospital program:

* In case of refusal or impossibility of the day hospital program: multidisciplinary follow-up "as usual" at the consultation center (outpatient group).
* In case of acceptance of the day hospital program (day hospital group): scheduling of 10 to 12 sessions over 12 weeks during a program session, followed by a new evaluation at the end of the program. Outpatient follow-up thereafter.

Outpatient follow-up consists of appointments with the psychiatrist, pediatrician, and dietitian, on average, every month.

Follow-up visits:

* Day hospital group only - at approximately 12 weeks: Visit 1bis: clinical evaluation at the end of the program + semi-structured interviews with parents
* Visit 2 - at 6 months: evaluations, with a search for clinical events + semi-structured interview with patients (either at V2 or V3)
* Visit 3 - at 12 months: evaluations, with a search for clinical events + semi-structured interview with patients (either at V2 or V3)

End of research visit:

- Visit 4 - at 5 years: evaluations, with a search for clinical events

Visits V2, V3, and V4 can be conducted by phone. Visit V4, not necessarily planned as part of the adolescent's follow-up, may be added to care if necessary. It can be conducted by phone, depending on the adolescent's choice.

For participants who have taken part in the day hospital program or outpatient follow-up before the implementation of this protocol and who meet the inclusion criteria, the information sheet will be provided to them during a consultation by an investigator, and non-opposition will be obtained at the next consultation. In case of agreement to participate, data from already conducted visits will be collected retrospectively, and patients will then be contacted for the yet-to-be-performed assessment visits at 6 months (if applicable), 1 year (if applicable), and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents in the age range of 12-18 years and their parents,
* First-time consultation at the MDA for anorexia nervosa (according to DSM-5) evolving for less than 12 months,
* Adolescents with clinical characteristics suitable for DH care.

Exclusion Criteria:

* Parents and/or children who do not speak French or cannot read or write,
* Patients who have been followed by an eating disorder specialist in the past 12 months (at the MDA or elsewhere) or previously hospitalized for anorexia nervosa,
* Patients who have undergone family therapy in the past,
* Patients with BMI less than 13 kg/m2 for those under 14 years old, or less than 14 kg/m2 for those over 14 years old at the initial assessment,
* Patients with a major psychiatric comorbidity or a metabolic condition interfering with eating or its regulation,
* Patients and families in a crisis situation requiring immediate hospitalization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients of any gender aged 12 to 18 years and their parents, seen in consultation for anorexia nervosa at the pedopsychiatric unit of the Cochin Hospital, Paris, France.
Sampling Method: Non-Probability Sample
Enrollment: 164 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of one or more clinical events | 1 year after inclusion
  Occurrence of one or more clinical events indicative of the progression of this disease (hospitalization, emergency room visits, major decompensation) at 1 year.
  Evaluate the impact of early intervention in DH on the clinical progression of the disease compared to the usual outpatient care.

SECONDARY OUTCOMES:
Occurrence of one or more clinical events | 5 years after inclusion
  Occurrence of one or more clinical events indicative of the progression of this disease (hospitalization, emergency room visits, major decompensation) at 5 years in both care groups.
  Evaluate the long-term impact of early intervention in DH on the clinical progression of the disease, compared to the usual outpatient care.
Conduct semi-structured qualitative interviews | After DH termination = 12 weeks after inclusion
  Conduct semi-structured qualitative interviews with parents after participation in the DH program.
  Explore the experience and perspectives of families participating in a new day hospital care program for adolescents with recent anorexia nervosa.
Satisfaction questionnaire CSQ-8 (Consumer satisfaction questionnaire) | After DH termination = 12 weeks after inclusion
  Satisfaction questionnaire at the end of DH care. Assess the satisfaction level of the patient and their parents regarding DH care.
  The range of possible scores is 8-32; (32 = higher satisfaction = better outcome, 8 = lower satisfaction)
Clinical characteristics collection | Inclusion
  Initial clinical characteristics at the time of inclusion. Determine predictive factors for the outcome at the end of the intervention and in the long term.
Socio-demographic characteristics collection | Inclusion
  Initial socio-demographic characteristics at the time of inclusion. Determine predictive factors for the outcome at the end of the intervention and in the long term.
Semi-structured interviews (DH program group) | From 6 to 12 months after the end of day hospital (visit 2 or 3 - DH program group)
  Semi-structured interviews 6 to 12 months after their discharge from day hospital (visit 2 or 3 - DH program group), to assess the impact on the evolution of symptomatology of the experience lived by adolescents in the care within the framework of this early management system for anorexia nervosa (HDJ group).

CONTACTS AND LOCATIONS:
Locations (1):
- Maison de Solenn Maison des Adolescents, Cochin Hospital, Paris, IDF, France

IPD SHARING:
Plan to Share IPD: Undecided